CLINICAL TRIAL: NCT06351670
Title: Personalised Monitoring of Early and Intermediate Age-related Macular Degeneration With Artificial Intelligence and Identification of Disease Progression in a Prospective, Multinational, Multicentre Observational Study
Brief Title: Personalised Monitoring of Early and Intermediate Age-related Macular Degeneration With Artificial Intelligence and Identification of Disease Progression
Acronym: SUDETES
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: University Medical Centre Ljubljana (Other); Centre Hospitalier Universitaire Dijon (Other); Queen's University, Belfast (Other); University of Zurich (Other); Vista Klinik (Other); Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Gregor Reiter, Principal Investigator, Medical University of Vienna
Other Study IDs: 1109/2024
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective, multinational, multicenter observational study is to to predict conversion of early and intermediate AMD with functional vision to advanced AMD with irreversible loss of vision on an individual-based level over 2 years. The main objectives of this study are:

* Identify and quantify focal and global alterations in the retina in regard to disease progression.
* Assess the individual risk of disease progression in intermediate AMD patients converting to advanced AMD based on imaging.
* Specify the course of disease in regard to the sequence of events that lead to the conversion to advanced AMD
* Enhance the ability to classify AMD using artificial intelligence in addition to traditional models.

All patients will be followed for 24 months with 6 month intervals to assess clinical changes. Monitoring of disease progression will be performed using the following routine in-vivo imaging procedures:

* Scanning Laser Fundus Photography
* Color Fundus Photography (CFP)
* Optical Coherence Tomography (OCT)
* Optical Coherence Tomography Angiography (OCTA) Patients will be asked for their medical history. Standard ophthalmic examination, as well as a questionnaire on visual function will be carried out.

No intervention will be performed during the study since no treatment is yet available within Europe. As soon as treatment is approved in the EU, patients in this cohort might receive treatment according to availability in their respective country and standard of care. If treatment will be performed, it will be as standard of care outside the study according to each country's standard of care and by EMA label.

ELIGIBILITY:
Inclusion Criteria:

* Age: 55-99 years old
* Early or intermediate AMD in at least one eye (drusen > 63 µm and/or any definite hyper- or hypopigmentary abnormalities with or without reticular pseudodrusen)
* If both eyes are eligible, both eyes will be included in the cohort study.
* Clear optical media and adequate pupillary dilation for imaging and functional testing.

Exclusion Criteria:

* Any surgical treatment of the eye within 3 months prior to baseline in the study eye
* History of anti-VEGF treatment in the study eye before baseline
* History of pseudophakic cystoid macular edema (Irvine Gass Syndrome) in the study eye
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure (IOP) ≥ 25 mmHg despite treatment with IOP lowering medication), or C/D Ratio > 0.9
* Any concurrent intraocular condition in the study eye (e.g. advanced cataract or moderate/severe diabetic retinopathy) that, in the opinion of the investigator, will most likely require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition
* Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could cause an unwanted effect on treatment efficacy, compliance or require intraocular surgery (except for cataract surgery and YAG capsulotomy) during the study period
* Presence of corneal decompensation, haze or scarring with an impact on BCVA
* Refractive error larger than 6 diopters. In case of pseudophakia or refractive surgery: History of refractive error larger than 6 diopters.
* Intake of drugs known to cause retinal toxicity (e.g. hydroxychloroquine or tamoxifen)
* Presence of active macular neovascularization at baseline

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from each center's respective outpatient clinic and/or by referral from primary eye care (e.g. optometrist).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To characterise and quantify focal and global changes of the retina by retinal imaging to identify patients at risk for conversion to advanced AMD. | 2 years
  The correlation between biomarkers (independent variables) and progression will be assessed by linear mixed models or prospectively by Cox-regression models.
  Artificial intelligence models will be applied to assess progression speed and predict local and global progression.
  Mixed Effects models will be calculated to estimate the association between independent variables, including the timepoint as an independent variable, on individual markers of progression (PR thinning and PR loss expansion).

SECONDARY OUTCOMES:
To identify and quantify disease progression-related biomarkers | 2 years
  Longitudinal assessments of imaging biomarkers are performed in a descriptive manner. The following biomarkers will be evaluated in detail as independent variables:
  * Drusen volume/Refractile drusen (scale, nl)
  * Subretinal Drusenoid Deposits (SDD) (scale, mm2)
  * Hyperreflective Foci (HRF) (scale, nl)
  * Thinning of outer retinal layers (PR thinning) (scale, µm)
  * Loss of outer retinal layers (RPE and PR) (scale, mm2)
  * PR loss/RPE loss ratio (scale, ratio)
  * Other retinal biomarkers if relevant to the progression of intermediate AMD to advanced AMD
  The correlation between biomarkers (independent variables) and disease progression will be assessed by linear mixed models or prospectively by Cox-regression models. Mixed Effects models will be calculated to estimate the association between independent variables, including the timepoint as an independent variable, on individual markers of progression (PR thinning and PR loss expansion).
To evaluate monitoring of AMD progression assisted by AI algorithms | 2 years
  The following will be provided by AI-based image analysis of the GA Monitor (independent variables used to detect an event for the Cox-regression model):
  * RPE integrity loss (mm2) in the 1mm central area, 6mm area, and the respective relative change to previous visit
  * PR integrity loss (mm2) in the 1mm central area, 6mm area, and the respective relative change to previous visit
  The following will be provided by AI-based image analysis of the Fluid Monitor (independent variables used to detect an event for the Cox-regression model):
  * Intraretinal fluid volume (nl) in the 1mm central area, 6 mm area, and the respective relative change to previous visit
  * Subretinal fluid volume (nl) in the 1mm central area, 6 mm area, and the respective relative change to previous visit
  * Pigment epithelium detachment volume (nl) in the 1mm central area, 6mm area, and the respective relative change to previous visit

CONTACTS AND LOCATIONS:
Locations (7):
- Medical University of Vienna, Vienna, Austria
- CHU Dijon, Dijon, France
- University Medical Center Ljubljana, Ljubljana, Slovenia
- Fundacio de Recerca Clinic Barcelona-Institut D Investigacions Biomed, Barcelona, Spain
- Switzerland (2):
  - Vista Klinik Binningen, Binningen
  - University of Zürich, Zurich
- Queen's Unviversity Belfast, Belfast, United Kingdom